CLINICAL TRIAL: NCT05677555
Title: Colchicine Influence on Chronic Inflammation in Hemodialysis Patients
Brief Title: Colchicine and Inflammation in Hemodialysis Patients
Acronym: CICI-HP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, ilia beberashvili MD, head of dialysis department, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9922
Record Dates: First submitted 2022-09-10; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: End Stage Renal Disease on Dialysis
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- colchicine group (Experimental): Treatment with colchicine 0.5 mg
  Interventions: Drug: Colchicine 0.5 MG
- placebo group (Placebo Comparator): Treatment with matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 MG — A total of 25 subjects will be randomized to treatment with COLCHICINE 0.5 mg, three times a week (at the end of each hemodialysis session) over the 3 month study period.
  Arms: colchicine group
Drug: Placebo — A total of 25 subjects will be randomized to treatment with matched placebo, three times a week (at the end of each hemodialysis session) over the 3 month study period.
  Arms: placebo group

SUMMARY:
Chronic, low-grade inflammation is regarded as a common comorbid condition in chronic dialysis patients.

Increased inflammatory markers in chronic dialysis patients are associated with adverse clinical outcomes .

Considering the association of low-grade inflammation with high rate of morbidity and mortality we decided to evaluate the anti inflammatory effect of colchicine on inflammatory markers in hemodialysis patients

DETAILED DESCRIPTION:
Adult end-stage kidney disease (ESKD) patients undergoing maintenance hemodialysis (MHD) experience high mortality and morbidity with diminished quality of life . Death and hospitalization rates in MHD patients correlate strongly with indicators of chronic inflammation .

Chronic, low-grade inflammation is regarded as a common comorbid condition in CKD, and particularly in chronic dialysis patients.Several circulating markers are commonly assessed as indicators of systemic inflammation. IL-1 is a pro-inflammatory mediator of both acute and chronic inflammation, and induces synthesis and expression of hundreds of secondary inflammatory mediators .IL-1β is the main form of circulating IL-1 and is initially synthesized as a precursor (pro-IL-1β) that becomes activated in the setting of a macromolecular structure known as the inflammasome , which is activated in CKD and perpetuates the inflammatory response .IL-6 is a pro-inflammatory cytokine that promotes inflammatory events through activation and proliferation of lymphocytes, differentiation of B cells, leukocyte recruitment, and induction of the acute-phase protein response in the liver .IL-6 can be induced by IL-1 and by TNF-α, the latter of which is a soluble receptor primarily produced by monocytes and macrophages and elevated in states of chronic inflammation .CRP is an acute phase reactant, downstream from IL-6, and is a more specific marker of plaque vulnerability and risk of cardiovascular events, with data suggesting it may play a direct role in atherogenesis rather than simply acting as a marker, as previously believed .

Increased inflammatory markers in chronic dialysis patients are associated with adverse clinical outcomes including all-cause mortality, cardiovascular events ,protein energy wasting and diminished motor function, cognitive impairment ,as well as other adverse consequences including CKD-mineral and bone disorder (CKD-MBD) ,anemia ,and insulin resistance .

Despite the strong evidence that the prevalence of chronic inflammation is high and it independently predicts numerous adverse clinical outcomes in chronic dialysis patients, the evidence for a role of inflammation in affecting outcomes is limited by the fact that most of the available evidence is epidemiological in nature, with some additional support provided by mechanistic animal studies .Strategies shown to reduce systemic inflammatory markers in chronic kidney disease and/or chronic dialysis patients include pharmacological and non-pharmacological approaches. Pharmacological strategies that have been evaluated are specific anti-cytokine therapies (anakinra, as well as IL-6 monoclonal antibody etc.), as well as non-specific agents with anti-inflammatory properties, including statins, angiotensin converting enzyme inhibitors and angiotensin receptor blockers, cholecalciferol (vit D), sevelamer, peroxisome proliferator-activated receptor-γ (PPAR-γ) agonists, and growth hormone .However, the data that reducing systemic inflammation improves clinical outcomes are currently lacking; this area represents an important future research direction.

Colchicine is an ancient medication that is currently approved for the treatment of gout and FMF .However, colchicine has a wide range of anti-inflammatory activities, and studies indicate that it may be beneficial in a variety of other conditions .In this respect, attention should be paid to the recently published article that shows that colchicine at a dose of 0.5 mg daily led to a reduction of inflammation expressed by serum CRP levels and a significantly lower risk of ischemic cardiovascular events than placebo among patients with a recent myocardial infarction .Interestingly, although acute preprocedural administration of colchicine did not lower the risk of percutaneous coronary intervention (PCI)-related myocardial injury, it successfully attenuated the increase in interleukin-6 and high-sensitivity C-reactive protein concentrations after PCI when compared with placebo .Recently reported that short-term administration of low-dose colchicine significantly alleviated endothelial inflammation with reduction of serum CRP concentration in coronary artery disease patients .It was found that short-term colchicine therapy dramatically reduced the expression levels of IL-1β, IL-6 and IL-18 by blockade of nucleotide-binding oligomerization domain-like receptors, pyrin domain-containing 3 (NLRP3) inflammasome activation in acute coronary syndrome patients .

The only paper reported on the use of colchicine in dialysis patients is the report on the use of colchicine in peritoneal dialysis (PD) rats with encapsulating peritoneal sclerosis .There is no information in the literature on whether colchicine affects inflammation measures in dialysis patients. Given the high morbidity and mortality in MHD patients, targeting inflammation represents a potentially novel and attractive strategy if it can indeed be shown to improve their adverse outcomes.

Considering the association of low-grade inflammation with high rate of morbidity and mortality in MHD population and anti-inflammatory potential of colchicine on the other hand, we decided to conduct the Colchicine Influence on Chronic Inflammation in Hemodialysis Patients (CICI-HP) study to evaluate the effects of colchicine on inflammatory markers as well as its safety profile in MHD patients.

The study will be conducted as a 3-month, double-blind, parallel-group, placebo-controlled, single center study. The study population will include 50 ESKD patients receiving MHD treatment with different degrees of low-grade inflammation (defined as plasma CRP above 10 mg/L and below 100 mg/L). A total of 50 subjects will be randomized to treatment with either colchicine 0.5 mg three times a week (at the end of each hemodialysis session) or matching placebo. Both patients and investigators (including doctors, nurses and dietitians) will be blinded to group assignment. Randomization codes will conceal until end of trial . The randomization list and all study products will be provided by "Super Pharm Professional" laboratory Petah Tikva .

After meeting all inclusion criteria all study participants will be seen at 4 visits over the 3 month period. All visits will take place in connection with a regular dialysis session. At all study visits predialysis blood samples will be collected in a fasting state from each study patient. The dietary energy and protein intake will be calculated and normalized for ideal body weight according to the European Best Practice Guidelines by skilled dietitian. Dietitian records based on self-completed food diaries with continuous 3-day dietary histories (including a dialysis day, a weekend day and a non-dialysis day) will be used to calculate the dietary intake. The same dietitian will perform all anthropometric measurements and calculation of daily calorie and protein intake per diaries records. During the dialysis session SNAQ questionnaires for appetite assessment will be filled out. At study entry, each participant will be instructed how to work with questionnaires. All participants will also fill out the EQ-5D questionnaires on their own, or will be assisted by an independent person if the patient himself unable to complete questionnaire. Handgrip strength (HGS) will be measured in all patients using the non-dominant hand. The patients will undergo BIA at approximately 30-minutes postdialysis.

The study parameters will be: SNAQ (the simplified nutritional appetite questionnaire) for appetite assessment; daily energy and protein intake for dietary assessment; EQ-5D for health-related QoL assessment; biochemical nutritional markers (serum albumin, creatinine, transferrin, uric acid, lipid profile, IGF-1), appetite-regulating peptides (leptin, acyl-ghrelin, obestatin, NPY); inflammatory biochemical mediators (CRP, neutrophil-to-lymphocyte ratio, IL-6, and TNFα); handgrip strength as functional assessment of muscle mass; anthropometric parameters (body weight, BMI, skinfold thickness, mid arm circumference and mid arm circumference calculated); lean body mass, % fat mass, fat free mass, phase angle measured by BIA, malnutrition inflammation score, geriatric nutritional risk index (GNRI) and objective score of nutrition on dialysis (OSND) as quantitative assessment of nutritional status.

All patients will undergo regular hemodialysis via their vascular access 4-5 h 3-4 times per week at a blood flow rate 250-300 mL/min. Bicarbonate dialysate (30 mEq/L) at a dialysis solution flow rate of 500 mL/min will be used in all cases. All patients will use the same high flux dialyser membrane (biocompatible) with surface area of 1.8-2.2m2 and patients won't use re-used dialyzer membrane. The efficiency of the dialysis will be assessed based on the delivered dose of dialysis (Kt/Vurea) using a single-pool urea kinetic model. Protein equivalent of nitrogen appearance (nPNA), an indirect indicator of protein intake, will be calculated from serum urea levels using three-point method.

During the study period (from screening to the last follow up visit - about 3 months period) we will monitor all morbid events for all study patients. Specific causes of hospitalization (grouped as infectious causes, cardiac causes, vascular-access related causes, and other causes classified according to ICD-9 codes) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-90 years, on MHD hemodialysis treatment at least 3 months
* Stable and adequate hemodialysis treatment three months prior to participation in study as defined by Kt/V > 1.2 and/or hemodialysis performed 4 hours 3 times weekly
* Patients with serum CRP ≥ 10 mg/L
* Informed consent obtained before any trial-related activities

Exclusion Criteria:

* PermCath use as vascular access
* Any intake of colchicine for the last three months before recruitment
* Critical illness as defined by the need of respiratory or circulatory support
* Known or suspected allergy to colchicine
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using contraceptive methods
* Patients with active malignant disease or liver cirrhosis or Severe hepatic disease( defined as ALT or AST levels >3 times upper normal range)
* Actively symptomatic gastrointestinal bleeding and inflammatory bowel disease
* CRP level above 100 mg/L
* Patients on chronic treatment with steroids on doses > 10 mg/day Prednisone (or equivalent)
* Patients treated with immunosuppressive agents
* Patients receiving any of the following medications: Astemizole, Cisapride, Pimozide or Terfenadine.
* Patients suffering from -Acute vasculitis, Severe systemic infections, Severe Heart failure (NYHA class IV), or Mental incapacity
* Any condition judged by the investigator to interfere with trial participation or evaluation of results or to be potentially hazardous to the patient
* A significant history of alcohol, drug or solvent abuse
* History of schizophrenia, history of psychiatric hospitalization
* unwillingness or language barrier
* The receipt of any investigational drug within 1 month prior to initiating of this study
* Scheduled renal transplantation (fixed date)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Inflammation assessed by measuring blood levels of inflammatory biomarkers | 3 months
  Investigate the effect of colchicine on the level inflammation blood biomarkers (C- reactive protein -CRP, IL-6, TNF-a) of adult patients on maintenance hemodialysis (MHD)
Incidence of treatment emergent adverse events as assessed by routine clinical and blood tests monitoring | 3 months
  In each visit (every month) participants will be interview for every change in their clinical status including specific known adverse events of colchicine (such as diarrhea , neuropathy, fever, muscle weakness). moreover, blood tests will be drawn for complete blood count and chemistry. physical examination will be carried out at ehch visit.

SECONDARY OUTCOMES:
Nutritional score- VAS - visual analog scale | 3 months
  - above 48 millimeteres is considered a good score for accessing no feeling of hunger
Quality of life score-SF-36- "36 item short form survey" | 3 months
  score range 0-100 - higher scores indicate better health status ( score of 50 is a normative value)
Body composition by bioimpedance-lean body mass | 3 months
  measurement of lean body mass will be described by killograms units
NUTRITIONAL SCORE- ADAT- appetite and diet assessment tool | 3 MONTHS
  - 1- very good 2-good 3- fair 4- poor 5-very poor
NUTRITIONAL SCORE- OSND- objective score of nutrition on dialysis | 3 MONTHS
  normal score 28-32, intermediate malnutrion 24-27, 23 and lower- severe malnutrition
NUTRITIONAL SCORE-SNAQ- simplified nutritional appetite questionnaire - score | 3 MONTHS
  - score at or below 14 indicates significant risk of at least 5 % weight loss within 6 months
NUTRITIONAL SCORE-MIS- malnutrition inflammation score | 3 MONTHS
  - 0 is normal, 30-severe degree of malnutrition and inflammation
Quality of life score-ESAS- Edmonton Sympthom Assessemnt System | 3 months
  - score between 1-10 . 10 is worsth
Quality of life score-EQ-5D - EuroQual-5 D | 3 months
  score between 0-100 , 0 is the worth health status as percieved by the patient, 100 is the best health status as percieved by the patient
Body composition by bioimpedance- fat mass | 3 months
  measurement of fat mass will be described by killograms units
Body composition by bioimpedance-phase angle | 3 months
  measurement of phase angle will be described by the time difference between adjacent current and voltage peaks, divided by 180 degrees

CONTACTS AND LOCATIONS:
Overall Officials: ILIA beberashvili, Professor, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Asaf ha Rofeh, MC, Zrifin, Israel

IPD SHARING:
Plan to Share IPD: Yes
Except for personal identities , we will share data including baseline characteristics of the study population, results and statistics of primary and secondary outcomes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the end of study period (after the last follow up visit - about 3 months period), and for one year thereafter.